CLINICAL TRIAL: NCT05793034
Title: Analysis of Predictive Factors for Overall and Progression-free Survival After Neurosurgery for Atypical or Anaplastic Meningioma
Brief Title: Predictive Factors for Survival in Aggressive Meningiomas
Acronym: 23Men
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3459
Record Dates: First submitted 2023-02-23; First posted 2023-03-31 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Meningioma; Meningioma Atypical; Anaplastic Meningioma
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological biomarker assessment (Other): FFPE tumor tissue will be processed with a number of molecular biology techniques
  Interventions: Diagnostic Test: Biological biomarker assessment

INTERVENTIONS:
Diagnostic Test: Biological biomarker assessment — IHC, PCR, NGS, methylome

SUMMARY:
The investigators plan to collect clinical and molecular data, including ICH, PCR, NGS and methylome, from patients operated on for grade 2 or grade 3 meningioma. The purpose of the study is to identify reliable and easy-to-assess predictive factors for recurrence and survival after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patient operated for atypical (grade 2) meningioma; or
2. Patient operated for anaplastic (grade 3) meningioma;
3. Timeframe for surgery, 1999-2019

Exclusion criteria

1) Patient lost at follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2026-01-07 (Estimated); Study Completion 2027-01-07 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) | 5 years on average
  Correlation from biomolecular data and RFS

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years on average
  Correlation from biomolecular data and OS

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy